CLINICAL TRIAL: NCT03565094
Title: Interventional, Open-label, Single- and Sequential-ascending-dose Study Investigating the Safety, Tolerability and Pharmacokinetic Profile of Lu AF28996 in Healthy Young Men
Brief Title: Single Dose of Lu AF28996 to Healthy Young Men
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: H. Lundbeck A/S (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17695A
Record Dates: First submitted 2018-06-08; First posted 2018-06-21 (Actual); Last update posted 2019-09-26 (Actual); Status verified 2019-09

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Lu AF28996 (Experimental): Lu AF28996 solution, cohort depending dose
  Part A:
  Cohort 1: single oral dose of Lu AF28996
  Cohorts 2-6: two single ascending oral doses of Lu AF28996 with a washout in between
  Possibility of 4 additional cohorts (Cohorts 7 to 10), allowing for the investigation of a potential 13 additional subjects
  Part B: 8 subjects (randomised to one of four treatment sequences)
  Interventions: Drug: Lu AF28996 solution; Drug: Lu AF28996 capsule

INTERVENTIONS:
Drug: Lu AF28996 solution — Oral solution (0.1-0.2 mg/mL)
  Following each cohort, a dosing conference will be held where tolerability, safety and preliminary PK results from the previous cohorts will be reviewed before deciding on the next doses
Drug: Lu AF28996 capsule — hard capsule orally QD: one dose lower than the highest dose level in part A

SUMMARY:
This study evaluates how increasing doses of Lu AF28996 enters, moves through and exits the body when given by mouth to healthy young men.

DETAILED DESCRIPTION:
Part A of the study consists of 6 groups (Cohorts 1 to 6) with 3 subjects in each, with the possibility of 4 additional cohorts. In cohort 1, the subjects will receive a single dose of Lu AF28996 by mouth. Following evaluation of data from the first dose, the subjects in the following cohorts are planned to receive two single increasing doses by mouth of Lu AF28996 on 2 separate days with a wash out (day or days without dosing) in between.

Part B is an open-label three-period crossover study in healthy young men to compare the PK of an oral capsule formulation with that of an oral solution formulation and to evaluate food effect following oral capsule administration of Lu AF28996.The subjects will be randomised to one of the four treatment sequences

ELIGIBILITY:
Inclusion Criterium:

Healthy, young, non-smoking men aged ≥18 and ≤45 years and with a body mass index (BMI) ≥18.5kg/m2 and ≤30kg/m2 at the Screening Visit

Other in- and exclusion criteria may apply

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 39 (Actual)
Dates: Start 2018-05-29 (Actual); Primary Completion 2019-08-17 (Actual); Study Completion 2019-08-21 (Actual)

PRIMARY OUTCOMES:
AUC 0-inf | From dosing to day 12 postdose
  area under the plasma concentration-time curve of Lu AF28996
Cmax | From dosing to day 12 postdose
  maximum observed plasma concentration of Lu AF28996
CL/F | From dosing to day 12 postdose
  Oral clearance of Lu AF28996

SECONDARY OUTCOMES:
Number of participants with Treatment-Emergent Adverse Events | From dosing to day 12 postdose
  Safety and Tolerability based on the safety assessments (clinical safety laboratory tests, vital signs, weight and ECG parameters)

CONTACTS AND LOCATIONS:
Overall Officials: Email contact via H. Lundbeck A/S, Study Director — LundbeckClinicalTrials@Lundbeck.com
Locations (1):
- QPS Netherlands BV, Groningen, Netherlands